CLINICAL TRIAL: NCT07233252
Title: Nephron-sparing Treatment Combining Tislelizumab and Nab-Paclitaxel for Renal Pelvic Cancer: An Open-Label, Single-Center, Single-Arm, Phase II Clinical Trial (TRUCE-U03)
Brief Title: Nephron-sparing Treatment of Tislelizumab + Nab-Paclitaxel for Renal Pelvic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRUCE-U03
Record Dates: First submitted 2025-08-09; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Renal Pelvic Carcinoma; Tislelizumab; PD-1 Inhibitor; Kidney-sparing; Nab-paclitaxel
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Arm1: Nab-Paclitaxel 125 mg/m2 IV on day 1 in combination with Tislelizumab 200mg IV on day 1 every 3 weeks for 2-3 cycles and then followed by efficacy evaluation. Patients achieved the criteria of "well response and tolerance" will undergo ureteroscopic biopsy. If residual lesions are detected under the ureteroscope, endoscopic intervention (e.g., laser ablation, cryoablation) should be carried out simultaneously to eliminate these residual lesions. Then, patients will receive no less than 2 cycles of maintenance therapy of Nab-Paclitaxel 125 mg/m2 IV on day 1 and Tislelizumab 200mg IV on day 1 every 3 weeks. Patients not achieved the criteria will be excluded from this study.
  Interventions: Drug: Nab-paclitaxel; Drug: Tislelizumab; Procedure: endoscopic intervention

INTERVENTIONS:
Drug: Nab-paclitaxel — Nab-Paclitaxel 125 mg/m2 IV will be administered on Day 1 every 3 weeks for 2-3 cycles before evaluation, then on Day 1 every 3 weeks for maintenance therapy after evaluation (only for patients who achieved the criteria of "well response and tolerance").
Drug: Tislelizumab — Tislelizumab 200mg iv will be administered on Day 1 every 3 weeks for 2-3 cycles before evaluation, then on Day 1 every 3 weeks for 3-6 cycles as maintenance therapy after evaluation (only for patients achieved the criteria of "well response and tolerance").
Procedure: endoscopic intervention — Patients who achieved the criteria of "well response and tolerance", but with residual lesions will receive endoscopic intervention (e.g., laser ablation, cryoablation) via ureteroscopy.

SUMMARY:
This study is designed as an open-label, single-arm, single-center, phase II clinical trial, aiming to evaluate the efficacy of nephron-sparing treatment combining Tislelizumab and Nab-Paclitaxel for HER-2 expressing renal pelvic cancer (RPC) . Patients enrolled will receive 2-3 cycles of Tislelizumab in combination with Nab-Paclitaxel every 3 weeks and then undergo evaluation. Patients who achieve all of the following criteria of "well response and tolerance" will receive further maintenance treatment:

(1)The patient achieves a complete response (CR) or partial response (PR) according to the RECIST 1.1 criteria, indicating that the tumor is well-controlled. (2) If the patient has residual lesions, it should be confirmed by the clinical physician that these lesions can be eliminated through laser ablation via ureteroscopy. (3)The patient has not experienced any treatment-related adverse events (TRAEs) that warrant discontinuation of therapy during systemic treatment. (4)The patient is willing to undergo further maintenance therapy. If the patient meets all the criteria above, ureteroscopic biopsy should be performed. If residual lesions are detected under the ureteroscope, endoscopic intervention (e.g., laser ablation, cryoablation) should be carried out simultaneously to eliminate these residual lesions. Patients who meet the above criteria will proceed with no less than 2 cycles of maintenance systemic therapy (Tislelizumab + Nab-Paclitaxel). Patients who do not meet the criteria will be excluded from the study and are recommended to undergo salvage radical nephroureterectomy (RNU) as soon as possible. One-year Nephron-Sparing Survival (1 year-NSS): Defined as the absence of surgical indications for nephrectomy due to progression or recurrence of upper urinary tract urothelial carcinoma, distant metastasis caused by the primary upper urinary tract tumor, or death from any cause within 1 year from the initiation of treatment. Treatment-related adverse events (TRAEs) will be recorded and evaluated according to CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged no less than 18 years old;
2. Suitable and planned to undergo laser ablation of renal pelvic tumors via ureteroscopy;
3. The tumor is located in the renal pelvis, diagnosed as upper tract urothelial carcinoma based on ureteroscopic biopsy, urinary cytology, or imaging examinations (CT, MRI, or PET-CT), without lymph node metastasis or distant metastasis, with a clinical stage of T1-2N0M0. Additionally, requiring maximum tumor diameter is less than 3 cm.
4. Expected survival time of more than 12 weeks;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2;
6. Agree to provide blood, urine, and tissue samples (for testing PD-L1 expression, HER-2, tumor mutation burden, etc.);
7. The organ function levels must meet the following requirements:

   Hematological indicators: Absolute neutrophil count ≥1.5×10^9/L, platelet count ≥80×10^9/L, hemoglobin ≥6.0 g/dL (can be maintained through symptomatic treatment); Liver function: Total bilirubin ≤1.5 times the upper limit of normal, alanine transaminase and aspartate transaminase ≤2.5 times the upper limit of normal; Renal function: Baseline ECT renography indicates a total renal glomerular filtration rate (GFR) ≥15 ml/min, with the affected-side GFR >10 ml/min, excluding the presence of a non-functional kidney (low-level decreasing curve on dynamic renal ECT imaging) on the affected side.
8. Participants are willing to join the study and be able to sign and comply the protocol.

Exclusion Criteria:

1. Concurrent primary malignancies in other sites are excluded, except for those with a history of other malignancies that have been treated and are currently stable.
2. Confirmed bilateral upper tract urothelial carcinoma (UTUC).
3. Presence of urothelial carcinoma in ureter or bladder is excluded, except for non-muscle-invasive bladder cancer that can be completely resected via transurethral resection of bladder tumor (TURBT).
4. Received a live attenuated vaccine within 4 weeks before treatment or plan to receive during the study period;
5. Active, known or suspected history of autoimmune disease;
6. Known history of primary immunodeficiency;
7. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
8. Pregnant or breastfeeding female patients;
9. Untreated acute or chronic active Hepatitis B or Hepatitis C infection. Patients receiving antiviral therapy may be eligible if viral load is under monitored, at the discretion of the physician based on the patient's individual condition;
10. Receiving immunosuppressive medication within 4 weeks prior to starting treatment, except nasal, inhaled, topical steroids, or systemic corticosteroids at physiological doses (i.e., not exceeding 10 mg/day of prednisone or equivalent dose of other corticosteroids);
11. Known or suspected allergy to Tislelizumab or Nab-Paclitaxel;
12. Active tuberculosis;
13. Previous treatment with PD-1/PD-L1/CTLA-4 immune checkpoint inhibitors or other immunotherapies;
14. Participation in another clinical study;
15. Fertile men or women without effective contraception;
16. Uncontrolled concurrent illness, including but not limited to:

(1)HIV infection (HIV antibodies positive); (2)Uncontrolled severe infection; (3)Uncontrolled systemic disease (such as severe psychiatric, neurological disorders, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver, or kidney disease, uncontrolled hypertension [i.e., hypertension of CTCAE grade 2 or higher despite treatment]); (4)Active hemorrhage or newly developed thrombotic disease. (5)Renal failure with CKD grade 5 and undergoing dialysis treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
One-year Nephron-Sparing Survival (1-year-NSS) | up to 1 year from the initiation of treatment.
  This is defined as the absence of surgical indications for nephrectomy due to progression or recurrence of upper urinary tract urothelial carcinoma, distant metastasis caused by the primary upper urinary tract tumor, or death from any cause within 1 year from the initiation of treatment. Kaplan-Meier curves will be constructed to provide descriptive information on nephron-sparing survival.

SECONDARY OUTCOMES:
Treatment-related adverse events (TRAEs) | From treatment initiation to 90 days after the last cycle of treatment.
  Treatment-related adverse events (TRAEs) ,defined as adverse events occurring from the start of treatment (C1D1) to 90 days after the completion of the last dose, including type, incidence rate, and severity grading (assessed according to the NCI-CTCAE V5.0 criteria)
Clinical Complete Response (cCR) | At the time of ureteroscopic biopsy (for efficacy evaluation) completed (within 14 weeks of the treatment initiated)
  Defined as the achievement of a complete response (CR) based on RECIST 1.1 criteria in radiological assessment following neoadjuvant therapy, negative results on urinary cytology, absence of residual tumor in the upper urinary tract as demonstrated by ureteroscopy, and no residual tumor in the specimen from ureteroscopic biopsy.
Objective Response (OR) | After completion of the last cycle (cycle 2 or cycle 3，each cycle is 21 days） of therapy.
  Defined as the achievement of partial response (PR) or complete response (CR) based on RECIST 1.1 criteria, as assessed by imaging studies at efficacy evaluation.
Events-Free Survival (EFS) | up to 5 years
  Defined as the time from treatment initiated to the first occurrence of delayed surgical disease progression, local tumor recurrence (including recurrence in the upper urinary tract and bladder, excluding non-muscle-invasive bladder cancer that can be resected by TURBT), distant metastasis, or death from any cause. The study will record the 1-, 2-, and 5-year EFS rates for the target population. Kaplan-Meier methods will be used to estimate the median EFS and 95% confidence interval limits, and Kaplan-Meier curves will be constructed to provide descriptive information on EFS
Overall Survival (OS) | up to 5 years
  Defined as the time from treatment initiated to death from any cause. The study will record the 1-, 2-, and 5-year OS rates for the target population. Kaplan-Meier methods will be used to estimate the median OS and 95% confidence interval limits, and Kaplan-Meier curves will be constructed to provide descriptive information on survival.
Recurrence-Free Survival (RFS) | up to 5 years
  Defined as the time from treatment initiated to the first occurrence of tumor recurrence (including recurrence in the upper urinary tract and bladder, excluding non-muscle-invasive bladder cancer that can be removed by TURBT). The study will record the 1-, 2-, and 5-year RFS rates for the target population. Kaplan-Meier methods will be used to estimate the median RFS and 95% confidence interval limits, and Kaplan-Meier curves will be constructed to provide descriptive information on RFS.
Cancer-Specific Survival (CSS) | up to 5 years
  Defined as the time from enrollment to death caused by the tumor. The study will record the 1-, 2-, and 5-year CSS rates for the target population. Kaplan-Meier methods will be used to estimate the median CSS and 95% confidence interval limits, and Kaplan-Meier curves will be constructed to provide descriptive information on CSS.

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Hu, PhD, Study Director — Tianjin Medical University Second Hospital
Locations (1):
- The Second Hospital of Tianjin Medical University, Tianjin, Outside U.S., China